CLINICAL TRIAL: NCT02978469
Title: Promoting Active Healthy Lifestyle of Adolescents With Brain Damage Due to Traumatic Brain Injury and Cerebral Palsy
Brief Title: Go For It: to Improve Levels of Daily Physical Activity and to Reduce the Sedentary Life Style of Adolescents With CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0082-15-ASF
Record Dates: First submitted 2016-11-17; First posted 2016-12-01 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: Habitual Physical Activity (HPA); Sedentary Behavior;
MeSH Terms: conditions — Cerebral Palsy; Phenylketonurias; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Life style changing: reducing sedentary behavior (Experimental): Meetings with social worker and physical therapist.
  Interventions: Other: Life style changing: reducing sedentary behavior
- Physical exercise group (Active Comparator): Physical therapy exercise training in group, strengthening and stretching muscles.
  Interventions: Other: Life style changing: reducing sedentary behavior

INTERVENTIONS:
Other: Life style changing: reducing sedentary behavior — The program includes 23 meetings held once per week (with holiday breaks). Each meeting lasts 90 minutes, consisting of exercise training.
  the group will meet for information providing and discussion. Participants are guided in the process of creating a focussed individualized activity plan.
  In the group setting they will experience a variety of activities enabling them to explore activities they prefer: each participant receive three personal consultation meetings. The group will experience sport and recreational activities with persons with physical impairments. Also activities in sport in community facilities.
  Other Names: 0082-15-ASF

SUMMARY:
Long hours of daily sitting and lack of Physical Activity (PA) are risk factors for morbidity and mortality.

People with movement disabilities, including adolescents with Cerebral Palsy (CP) tend to lead a sedentary life styl and have have poor physical fitness. Adolescents with CP where found to be inactive most of the day thus, they are in greater risk of disease than the general population. In addition, over the years, people with disabilities experience physical and functional deterioration. Reducing sedentary behavior and increasing daily activity can reduce health risk factors among the adolescents with CP, reduce secondary impairments and preserve function.

Interventions that included exercise alone has not resulted in physical activity and participating in a structured training did not continue after cessation intervention.

The objectives of this study are to establish effective programs aiming to promote an active life style among adolescents and young adults with CP and to evaluate there outcomes.

Specific objectives- Stage 1- Identifying barriers and facilitators for reducing sedentary behaviors and increasing physical activity among adolescents and young adults with CP. As well as, identifying mediators, needs and preferences for reducing sedentary behaviors and increasing physical activity among adolescents and young adults with CP.

Stage 2- Based on stage 1- Establishing an intervention for reducing sedentary behaviors and increasing physical activity among adolescents.

Stage 3- translating and developing questioners for the study.

* Translating the ASK-Performance and the ASK-Capability questionnaires to Hebrew and validating the Hebrew translation.
* Developing a self-efficacy perception questioner for increasing physical activity and reducing and sedentary behavior.
* Translating to Hebrew, adjusting and validating an activity diary.

Stage 4- evaluating the effectiveness of the proposed intervention program on reducing sedentary behaviors and increasing physical activity among adolescents and young adults with CP.

DETAILED DESCRIPTION:
Stage 1 focus group- Identifying barriers and facilitators for reducing sedentary behaviors and increasing physical activity as well as, identifying mediators, needs and preferences for reducing sedentary behaviors and increasing physical activity.

Stage 2- Based on stage 1- Establishing an intervention for reducing sedentary behaviors and increasing physical activity among adolescents. The intervention group will receive behavior-modification in group. The control group will get physical exercises.Stage 3- translating and developing questioners for the study.

* Translating the ASK-Performance and the ASK-Capability questionnaires to Hebrew and validating the Hebrew translation.
* Developing a self-efficacy perception questioner for increasing physical activity and reducing and sedentary behavior.
* Translating to Hebrew, adjusting and validating an activity diary.

Stage 4- evaluating the effectiveness of the proposed intervention program on reducing sedentary behaviors and increasing physical activity among adolescents and young adults with CP. The outcome measures will measure change from base line after intervention and 4-6 months after intervention finished.

All partners of this project will obtain approval for experiments on human subjects from their local committees. Each subject (or parents/guardians for the participation of minor subjects) will be able to sign an informed voluntary consent form, consistent with the Helsinki Declaration, after reading a detailed explanation and having an oral Q/A session with the investigator.

Recruitment: Prospective focused direct mailing or personal contacts will be initiated with the parents/guardians of children with CP who are ambulatory, who had been seen by physiotherapists in social groups and schools.

Inclusion exclusion criteria for Focus Groups:

* 30 adolescents with Cerebral Palsy
* aged 14-25yrs
* mobility level GMFCS I, II & III and
* 20 Typically Developed individuals same age group
* with verbal ability suitable for discussion
* Cognitive level sufficient to comprehend and cooperate with measurements.
* Parent or the individual (if above 18) has agreed to participate in the study

Exclusion criteria:

* Unstable medical situation
* Progressive degenerative condition of the Central Nervous System (CNS) or musculoskeletal system.

Inclusion exclusion criteria for intervention groups:

* adolescents and young adults with bilateral spastic CP
* at GMFCS level I, II and III
* age 14-25 yrs
* can speak their native language fluently
* are able to follow verbal instructions
* are willing to train in a group.

The exclusion criteria:

adolescents and young adults who had orthopedic surgery or tone reduction interventions (e.g. botulinum toxin injections, history of baclofen pump or selective dorsal rhizotomy) within 6 months prior to this study

- have exercise induced asthma or cardiac problems.

Inclusion criteria for validation ASK & Self Efficiency Questionnaire study:

* 30 Children and adolescents with CP
* age 5-20yrs
* GMFCS I;II;III.
* Cognitive level sufficient to comprehend and cooperate with measurements.
* Parent or the subject (if above 18) has agreed to participate in the study

Exclusion criteria:

* Unstable medical situation
* Progressive degenerative condition of the CNS or musculoskeletal system

Outcome measurements:

1. Habitual Physical Activity (HPA).Physical activity is recorded using an "ActivPAL3™" (PAL Technologies, Glasgow, UK) tri-axial accelerometer-based activity monitor.
2. 6 min walk test (6minWT): This test measures the self-paced distance in meters walked in 6 minutes on a flat, firm surface.
3. 10 meter walk test (10MWT): This self-paced test measures gait speed, important for safe community mobility (e.g., crossing streets in response to signals).
4. Timed Up-and-Go (TUG): This test measures mobility for those able to walk on their own (assistive device permitted).
5. Functional Mobility Scale (FMS): The FMS uses three distances (5, 50 and 500m) which represent typical distances walked by children at home, at school, and in the wider community.
6. The Activities Scale for Kids (ASK) is a child self-report measure of physical disability. It is designed for children five to 15 years of age who are experiencing limitations in physical activity due to musculoskeletal disorders.
7. The Pediatric Evaluation of Disability Inventory™ Computer Adaptive Test (PEDI-CAT) measures abilities in the three functional domains of Daily Activities, Mobility and Social/Cognitive. The PEDI-CAT's Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex, multi-step life tasks.
8. Self efficiency questionnaire: for evaluating perception of self efficiency for engaging in physical activity and reducing sedentary behavior.

Statistics:

Focus group: Coding text and theorizing: In grounded theory research. Identifying anchors that allow the key points of the data to be gathered. Collections of codes of similar content that allows the data to be grouped.

Repeated measures analysis of variance (ANOVA) will be used to determine the effects and compare the two groups methods.

A correlation test will take place between the ASK Capability and the PEDI-CAT. A correlation test will take place between the ASK PERFORMANCE and the results from the accelerometers.

One-way ANOVA test by separation the sample to severity groups, according to the GMFCS levels, using the age as a co-variant.

ELIGIBILITY:
Inclusion Criteria:

Intervention group:

* children, adolescents and young adults age 14-25 yrs
* with bilateral spastic Cerebral Palsy
* at GMFCS level I, II and III
* can speak their native language fluently
* able to follow verbal instructions
* willing to train in a group.

For ASK: age 5-18yrs.

* children, adolescents and young adults age 5-18yrs
* with bilateral spastic Cerebral Palsy
* at GMFCS level I, II and III
* can speak their native language
* able to follow verbal instructions

The exclusion criteria:

* Individual who had orthopedic surgery or tone reduction interventions (e.g. botulinum toxin injections, or have a history of baclofen pump or selective dorsal rhizotomy within 6 months prior to this study
* have exercise induced asthma or cardiac problems.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
an ActivPAL3™ (PAL Technologies, Glasgow, UK) tri-axial accelerometer-based activity monitor. | Measuring changes: Base line: time 1 before intervention. time 2: changes immediately after finish intervention. time 3: changes 6 months after time 2.
  tri-axial accelerometer-based activity monitor. ActivePal accelerometer, is currently considered a reference method for discriminating sitting, standing, and ambulation.

SECONDARY OUTCOMES:
6minWT | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention. time 3: 6 months after time 2.
  6 min walk test (6minWT): This test measures the self-paced distance in meters walked in 6 minutes on a flat, firm surface. This test assesses the sub-maximal level of functional capacity where most activities of daily living are performed and therefore reflects the effort required for daily physical activities.
10MWT | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention. time 3: 6 months after time 2.
  10 meter walk test (10MWT): This self-paced test measures gait speed, important for safe community mobility (e.g., crossing streets in response to signals). The 10MWT is measured by the time required to walk 10 m. It is a short and convenient test that can be applied to any subject able to ambulate that distance. A variation is the time to walk 10 m as fast as possible.
TUG | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention. time 3: 6 months after time 2.
  Timed Up-and-Go (TUG): This test measures mobility for those able to walk on their own (assistive device permitted). The test includes standing up from a chair, walking 3 m, turning 180°, walking back to the chair and sitting down. The test is measured by the total time to complete the task.
FMS | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention. time 3: 6 months after time 2.
  Functional Mobility Scale (FMS): The FMS uses three distances (5, 50 and 500m) which represent typical distances walked by children at home, at school, and in the wider community. For each distance, a rating of 1 to 6 was assigned, depending on the amount of assistance required for mobility. The rating is performed according to child/parent report of what the child does and is not by clinical observation.
ASK | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention. time 3: 6 months after time 2.
  The Activities Scale for Kids is a child self-report measure of physical disability. It is designed for children five to 15 years of age who are experiencing limitations in physical activity due to musculoskeletal disorders.
PEDI-CAT | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention, 4 months after starting intervention.
  The PEDI-CAT measures abilities in the three functional domains of Daily Activities, Mobility and Social/Cognitive.
Self efficiency questionnaire | Measuring changes on time line: Base line: time 1 before intervention. time 2: immediately after finish intervention. 4 months after starting intervention.
  Physical activity and sedentary behavior self efficiency questionnaire. include 17 facets 4 choices of agreements with statements.

CONTACTS AND LOCATIONS:
Overall Officials: Leonel Copeliovitch, MD, Principal Investigator — Human Motion Analysis Laboratory, Assaf Harofe Medical Center Zerifin Israel

IPD SHARING:
Plan to Share IPD: No